CLINICAL TRIAL: NCT01479634
Title: Early Antiretroviral Therapy in Resource Limited Settings in Patients With High CD4+ Cell Counts (EARLI)
Brief Title: Early HIV Therapy in Patients With High CD4 Cell Counts
Acronym: EARLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University Joint AIDS Program (Other); Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARLI
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: HIV; ART
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Treatment for HIV in participants with CD4+ cell counts 250-350 cells/uL
  Interventions: Drug: Standard ART
- Arm B (Active Comparator): Treatment for HIV in participants with CD4+ cell counts >350 cells/uL
  Interventions: Drug: Study-Provided ART

INTERVENTIONS:
Drug: Standard ART — Standard Ugandan 3-drug antiretroviral therapy regimen consistent with current practices
  Arms: Arm A
Drug: Study-Provided ART — Study provided drugs:
  1. Truvada® (one tablet PO daily of fixed dose combination consisting of tenofovir disoproxyl fumarate [TDF] and emtricitabine [FTC]) PLUS
  2. Efavirenz [EFV]
  Other Names: 1) FTC/TDF; 2) Sustiva®
  Arms: Arm B

SUMMARY:
A study of antiretroviral therapy (ART) initiation under a "streamlined model of care" in HIV-positive patients with CD4+ cell counts greater ≥ 250 cells/uL

DETAILED DESCRIPTION:
After dramatic progress in recent years, HIV care for patients in resource limited settings is rapidly evolving to newer models of care delivery. Governments, non-governmental organizations and charitable foundations are placing increasing scrutiny on the programmatic costs associated with delivering antiretroviral therapy (ART). Given these realities, if the global ART roll-out is to continue successfully, we must develop innovative new ways of providing HIV care and ART that are more efficient, more cost-effective, and tightly integrated within country-level health systems. We must treat more patients with fewer resources, and we need sustainable simple models for ART delivery.

These goals can be accomplished building on several existing knowledge points. First, initiating ART at earlier disease stages and at higher CD4+ cell counts may prevent irreversible immunologic damage, prevent opportunistic infections and non-AIDS-associated morbidities, and may prevent death. International and national HIV policy bodies have increasingly recognized this and adjusted recommendations in this direction. Second, ART initiation at higher CD4+ cell counts is less complex, triggers fewer complications, and is less costly to healthcare systems. Third, patients responding to therapy and doing well require fewer physician-administered follow-up visits. This can allow for "task-shifting" to non-MD providers, and the establishment of tiered healthcare delivery down the spectrum of medical acuity. Fourth, the lack of viral load monitoring is responsible for major structural problems in how we deliver ART, causing delays in recognizing ART failure, preventing clinicians from diagnosing HIV drug resistance, and making the decision to switch a patient to a new ART regimen very error-prone.

The EARLI study is a pilot study that will address and investigate all of the above critical issues. This study will focus exclusively on asymptomatic patients with CD4 cell counts ≥250 cells/uL. These relatively healthier individuals are well suited to a more streamlined approach to ART delivery and healthcare provision.

Primary Objectives:

A. To evaluate the 48 week efficacy of ART initiated in asymptomatic individuals with high CD4+ cell counts (CD4+ > 250 cells/uL) and provided in a "streamlined" mode of care.

B. To evaluate the programmatic costs of streamlined ART delivery to asymptomatic high CD4+ count individuals.

Secondary Objectives:

A. To evaluate the 96 week efficacy of ART initiated in high CD4+ cell count individuals.

B. To identify predictors of retention in care among high CD4+ cell count ART initiators.

C. To assess adverse events among high CD4+ cell count ART initiators.

D. To assess medication adherence among high CD4+ cell count ART initiators.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection diagnosed by a rapid HIV test or any licensed ELISA test kit and documented in the participant's medical chart and re-verified at the time of study screening (hereafter: "screen date").
* Most recent CD4+ cell count ≥ 250 cells/uL:

Arm A: CD4+ cell count 250-350 cells/uL Arm B: CD4+ cell count >350 cells/uL

* Age ≥ 18 years.
* Residence within a 30 kilometer radius of the Bwizibwera HC-IV.
* Willing to initiate ART if the CD4+ cell count is ≥ 350 cells/uL.
* The following laboratory values obtained at the screening visit:

  * Absolute neutrophil count (ANC) ≥ 500 cells/uL
  * Hemoglobin ≥ 7.0 g/dL
  * Platelet count ≥ 50,000/uL
  * ALT (SGPT) ≤ 5 times greater than the upper limit of normal
  * Estimated glomerular filtration rate (eGFR) of ≥ 60 mL/minute by the Modification of Diet in Renal Disease (MDRD) formula:

eGFR = 186 * Serum creatinine-1.154 * Age-0.203 * [1.21 if African] * [0.742 if female]

* Ability to swallow oral medications.
* Ability and willingness of participant to give informed written consent.

Exclusion Criteria:

* Receipt at any time prior to study entry of > 7 days cumulative treatment with any ARV or combination of ARVs, except ARVs taken for any length of time during pregnancy for the prevention of mother to child transmission (pMTCT) or ARVs taken for occupational exposure.
* For Arm B participants only: allergy/sensitivity to TDF, FTC, EFV, RTV, LPV or formulations of any of these three medications, or to co-formulated Truvada®.
* Active World Health Organization (WHO) HIV stage 3 or 4 illness
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
48-Week Efficacy | When all participants reach 48 weeks on study
  Proportion of patients with virologic suppression (HIV-1 plasma RNA ≤400 copies/cc) at 48 weeks, stratified by study arm.
Programmatic Costs | When all participants reach 48 weeks on study
  Total estimated costs of provider time, medications, diagnostic testing, and healthcare facility infrastructure per patient treated with ART for one year, stratified by study arm

SECONDARY OUTCOMES:
96-Week and 144-Week Efficacy | When all particiants reach 96 and 144 weeks on study, respectively
  Proportion of patients with virologic suppression (HIV-1 plasma RNA ≤400 copies/cc) at 96 and 144 weeks, stratified by study arm.
Predictors of Retention in Care | When all participants reach 48 weeks on study, then again 144 weeks on study
  Factors statistically significantly associated with attendance at all scheduled clinical visits throughout the first 48 weeks of ART, and throughout the full 144 week study period, stratified by study arm.
Adverse Event Rates | When all participants reach 48 weeks on study, then again at 144 weeks
  Describe grade 3 or 4 toxicities (defined by NIH DAIDS scale) that occur throughout the first 48 weeks of ART, and throughout the full 144 week study period, stratified by study arm. These will be assessed by active and passive ascertainment and clinical verification, stratified by study arm.
Medication Adherence | When all participants reach 48 weeks on study
  Proportion of total medication doses taken by patients at 48 weeks, assessed by pharmacy refill records, stratified by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Study Chair — University of California, San Francisco, San Francisco, CA, USA; Vivek Jain, MD, Principal Investigator — University of California, San Francisco, San Francisco, CA, USA; Moses Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University School of Medicine, Kampala, Uganda
Locations (1):
- Bwizibwera Level IV Health Center, Bwizibwera, Mbarara district, Uganda

REFERENCES:
- [Result] Jain V, Byonanebye DM, Amanyire G, Kwarisiima D, Black D, Kabami J, Chamie G, Clark TD, Rooney JF, Charlebois ED, Kamya MR, Havlir DV; SEARCH Collaboration. Successful antiretroviral therapy delivery and retention in care among asymptomatic individuals with high CD4+ T-cell counts above 350 cells/mul in rural Uganda. AIDS. 2014 Sep 24;28(15):2241-9. doi: 10.1097/QAD.0000000000000401. PMID 25022596
- [Derived] Jain V, Chang W, Byonanebye DM, Owaraganise A, Twinomuhwezi E, Amanyire G, Black D, Marseille E, Kamya MR, Havlir DV, Kahn JG. Estimated Costs for Delivery of HIV Antiretroviral Therapy to Individuals with CD4+ T-Cell Counts >350 cells/uL in Rural Uganda. PLoS One. 2015 Dec 3;10(12):e0143433. doi: 10.1371/journal.pone.0143433. eCollection 2015. PMID 26632823
- See also: MU-UCSF Research Collaboration website — http://www.muucsf.org/